CLINICAL TRIAL: NCT05845684
Title: Yenidoğan yoğun bakımda Uygulanan Fizyoterapi programının prematüre Bebeklerin Motor ve Beslenme performansına Etkisi
Brief Title: The Effect of the Physiotherapy Program Applied in the Neonatal Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Nilay Comuk Balci, Pt, Phd, Assoc. Prof., Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021/608
Record Dates: First submitted 2023-04-26; First posted 2023-05-06 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Premature; Infant, Light-for-dates; Neonatal Disease; Neurodevelopmental Disorders; Motor Delay
MeSH Terms: conditions — Premature Birth; Infant, Newborn, Diseases; Neurodevelopmental Disorders; Psychomotor Disorders | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trial group (Experimental): The physiotherapy group will receive a 10-minute massage in 30-minute sessions, 3 days a week for 1 month, oral and intraoral tactile stimulations, and non-nutritive sucking exercises to stimulate sucking. Positioning will be done for 15 minutes for mobilization purposes.
  Interventions: Other: Physiotherapy application
- control group (Other): In the control group, daily standard care practices will be performed.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Physiotherapy application — massage, oral and intraoral tactile stimuli and non-nutritive sucking will be performed to stimulate sucking, and massage applications and neurodevelopmental therapy for motor development.
  Arms: trial group
Other: Control Group — standard daily applications will be performed on patients
  Arms: control group

SUMMARY:
The aim of our study is to examine the effects of the physiotherapy program applied in the NICU on motor performance, behavior, transition time to full enteral feeding, and feeding performance in preterm infants.

DETAILED DESCRIPTION:
Preterm babies have to stay in neonatal intensive care units (NICU) because they cannot complete intrauterine development and have difficulty maintaining their vital functions.

In very low birth weight babies, feeding may not be started at the desired time due to medical problems. Total parenteral nutrition should be started in order to prevent growth retardation in the baby who cannot receive adequate enteral nutrition in the first days. The infant who tolerates enteral feeding should also be transitioned to full enteral feeding as soon as possible. Early enteral nutrition and intensive early parenteral nutrition reduce growth retardation and improve the infant's mental developmental scores. The frequent occurrence of feeding intolerance in preterm infants with very low birth weight, especially extremely low birth weight, and the risk of NEC, which is a serious cause of mortality and morbidity in these infants, prevent reaching the desired nutritional goals. Therefore, the optimum initiation time and rate of increase of enteral feeding are still uncertain for these infants. The main purpose of preterm nutrition should be to minimize the problems that may occur in the short and long term. The aim of our study is to examine the effects of the physiotherapy program applied in the NICU on motor performance, behavior, transition time to full enteral feeding and feeding performance in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Born 30 weeks or younger of gestational age, Body weight below 1500 g, The baby's vital signs are stable.

Exclusion Criteria:

* Infants undergo surgery, Taking antibiotics or phototherapy, Having a genetic syndrome • Having other medical conditions that may affect physiotherapy practices, such as multiple congenital anomalies, tracheoesophageal fistula, diaphragmatic hernia, congenital heart malformation, and/or necrotizing enterocolitis, The baby is intubated.

Ages: 10 Days to 20 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-12-31 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Dubowitz Neurological Assessment | 10 minutes
  Neurological assessment of the newborn infant.
Preterm Oral Feeding Readiness Assessment Scale | 10 minutes
  preterm infant oral feeding readiness instrument consisting of items in relation to corrected gestational age, behavioral state, global posture and tone, gag reflex, tongue movement and cupping, jaw movements and maintenance of an alert state

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Comuk Balci, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Nilay Çömük Balci, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Comuk Balci N, Takci S, Seren HC. Improving feeding skills and transition to breastfeeding in early preterm infants: a randomized controlled trial of oromotor intervention. Front Pediatr. 2023 Sep 18;11:1252254. doi: 10.3389/fped.2023.1252254. eCollection 2023. PMID 37790695